CLINICAL TRIAL: NCT02094287
Title: Placebo Effect in Atopic Dermatitis - Increase the Pharmacological Effect of Itching Caused by Classical Conditioning and Expectancy Processes: A Randomized Controlled Trial
Brief Title: Placebo Effect in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margitta Worm (Other)
Collaborators: University of Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Margitta Worm, Prof. Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PlacItch; 2008-008474-31 (EudraCT Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Dimethindene; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- verum, instruction, conditioning (Experimental): This group received dimetindene and instructions about dimetindene and its effectiveness. One classical conditioning process with saline was applied during the skin prick test procedures.
  Interventions: Drug: dimetindene; Behavioral: instruction; Other: conditioning
- verum, instruction, no conditioning (Experimental): This group received dimetindene and instructions about dimetindene and its effectiveness. No conditioning process were applied
  Interventions: Drug: dimetindene; Behavioral: instruction
- placebo, instruction, conditioning (Experimental): This group received a placebo (saline) as intravenously administered substance. But instructions about receiving dimetindene and its effectiveness were given. One classical conditioning process was applied during the skin prick test procedures.
  Interventions: Behavioral: instruction; Other: conditioning
- verum, no instruction, no conditioning (Experimental): Dimetindene was covertly administered (unawareness of treatment). No instruction and no conditioning were given.
  Interventions: Drug: dimetindene

INTERVENTIONS:
Drug: dimetindene — receiving either dimetindene or a placebo (saline) via infusion
  Arms: verum, instruction, conditioning; verum, instruction, no conditioning; verum, no instruction, no conditioning
Behavioral: instruction — information about the drug dimetindene and its efficacy versus no information and unawareness of treatment influencing expectations of an efficient treatment
  Arms: placebo, instruction, conditioning; verum, instruction, conditioning; verum, instruction, no conditioning
Other: conditioning — classical conditioning; experiencing and observing the efficiency of a drug manipulated by a conditioning process versus no learning experience.
  Other Names: learning experience
  Arms: placebo, instruction, conditioning; verum, instruction, conditioning

SUMMARY:
The study is initiated in the indication of atopic dermatitis to study the impact of placebo in the treatment of pruritus. Classical conditioning and expectation via instructions/anticipation maintain the effect of placebo.

ELIGIBILITY:
Inclusion Criteria:

* SCORAD-Score < 50 points
* basic experimental pruritus >= 3 points on a numeric rating scale
* no acute eczema on their forearms
* no systemic treatments for skin diseases for at least four weeks
* no topical treatment on their arms for at least two weeks

Exclusion Criteria:

* intake of antihistamines
* pregnancy and lactation
* serious dysfunctions of the liver, kidneys or thyroid
* prostatic hyperplasia
* patients with tumors, major cardiovascular diseases, immunosuppression
* glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the experimental pruritus intensity on a 10-point-rating scale between the groups | assessed over a time frame of 2 days
  The pruritus intensity is assessed at different time points during a time frame of 2 days. The results are compared between the groups.

SECONDARY OUTCOMES:
Change of the severity of atopic dermatitis (SCORAD) and comparison between the groups | assessed over a time frame of 2 days
  Change of SCORAD is assessed on day 1 and day 2.
Changes of Wheal sizes experimentally provoked by skin prick test. | assessed over a time frame of 2 days
  The changes of wheal sizes due to the administered intervention at different time point during a time frame of 2 day is assessed in square millimeters. The results are compared between the groups.
Changes of clinical, atopic itch intensity on a 10-point-rating scale | assessed over a time frame of 2 days
  Changes of clinical itch intensity assessed on day 1 and day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - University Medicine Berlin, Berlin
  - University of Hamburg, Hamburg